CLINICAL TRIAL: NCT04349865
Title: Assessment of LRRK2 Activity in G2385R Carriers and Markers Predicting Conversion to and Progression of Parkinson's Disease
Brief Title: LRRK2 Activity and Markers of Parkinson's Disease in G2385R Carriers
Status: Completed | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Principal Investigator, Piu Chan, Principal Investigator, Xuanwu Hospital, Beijing
Other Study IDs: LRRK2G2385R
Record Dates: First submitted 2020-01-18; First posted 2020-04-16 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Parkinson Disease
Keywords: LRRK2 G2385R variant; Parkinson's disease; LRRK2 activity
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — venous blood collected with EDTA anticoagulant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Idiopathic PD: PD patients without the LRRK2 G2385R mutation
- LRRK2 G2385R PD: PD patients with the LRRK2 G2385R mutation
- LRRK2 G2385R carriers: Subjects without PD who screen positive for the LRRK2 G2385R mutation
- Controls: Subjects without PD who screen negative for the LRRK2 G2385R mutation

SUMMARY:
The goals of this study are

1. To compare the functional effects of the LRRK2 G2385R variant among carriers with and without Parkinson's disease (PD) and non-carriers with and without PD
2. To investigate the relationship between functional effects of the LRRK2 G2385R variant and PD associated phenotype
3. To investigate the biomarkers associated with PD conversion in the LRRK2 G2385R variant carriers
4. To compare the immune-related differences between PD patients/unaffected individuals with and without the LRRK2 G2385R mutation, and to investigate the effects of immune dysfunction on the clinical expression of PD

DETAILED DESCRIPTION:
Pharmaceutical companies with LRRK2 kinase inhibitor programs are close to Phase 1 clinical testing. Phase II proof-of-concept clinical trials will need to be conducted in LRRK2 manifesting mutation carriers. This is currently a challenging task given the limited availability of this cohort.

While the LRRK2 G2019S mutation is the most common mutation present in Caucasians and certain ethic groups, the G2385R variant has been identified as a risk factor for sporadic PD in the Asian population (Chinese Han, Japanese and Korean). In fact, in these populations, the occurrence of this mutation is thought to be higher than (up to 4% of PD patients) the occurrence of the G2019S mutation in the Caucasian population. In contrast to G2019S, this variant has not been fully characterized. For example, there has been controversy regarding its kinase activity with some reporting higher and others lower activity. A systematic biochemical characterization of the G2385R is necessary to determine if this cohort may be useful in LRRK2 kinase inhibitor trials.

Although there were significant studies on the clinical characterization of LRRK2 risk variant carriers with or without PD, little is known which factor is more specific in predicting the conversion to PD and which biomarker can be used to measure the disease progression. Identifying these clinical phenotype and biomarkers will be critical for studying pharmaceuticals effective for PD.

Several lines of evidence point to a role of LRRK2 in the immune system. Particularly high LRRK2 expression has been discovered in macrophagic and monocytic cells, but not T-cells, leading to speculation of a functional role for LRRK2 in the innate immune system. LRRK2 is also expressed in toll-like receptor 4 (TLR-4)-activated microglia, brain-resident macrophage cells that have been implicated in the pathology of PD brain, and LRRK2 modulates proinflammatory responses in these cells via several immune signaling pathways. Moreover, enhanced neuroinflammation may contribute to neurodegeneration in PD patients carrying LRRK2 mutations. Further, recent genome-wide association studies highlight LRRK2 in the modification of susceptibility to the chronic autoimmune Crohn's disease and Mycobacterium leprae infection, raising the possibility that LRRK2 may contribute to PD through immunogenic mechanisms. Although neuroinflammation as a primary trigger or secondary process linked to PD remains unclear, the link between LRRK2 and the immune system provides an intriguing possibility for a potential pathogenic mechanism as well as aid in the identification of potential markers of LRRK2-related immune function that could inform therapeutic development and/or act as potential pharmacodynamic measures of LRRK2 activity.

This study will take advantage of the larger cohorts of LRRK2 G2385R variant carriers with or without PD established by the Chinese Parkinson Study Group in China.

ELIGIBILITY:
Inclusion Criteria:

1. PD patients:

   * A diagnosis of Parkinson's disease according to the 2015 MDS PD diagnostic criteria.
   * Willingness to take genetic testing.
2. Unaffected subjects:

   * Individuals aged 55 years or older without a diagnosis of PD.
   * Willingness to take genetic testing.

Exclusion Criteria:

□ Clinically significant neurological disorders.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: (1) PD patients are from the Chinese National Consortium of Parkinson Disease (CNCPD) cohort; meanwhile, new patients are enrolled from outpatient and inpatient departments.
  2) Unaffected subjects are from a large population-based cohort (the Beijing Longitudinal Study of Aging).
Sampling Method: Non-Probability Sample
Enrollment: 211 (Actual)
Dates: Start 2018-05-22 (Actual); Primary Completion 2020-12-25 (Actual); Study Completion 2020-12-25 (Actual)

PRIMARY OUTCOMES:
LRRK2 activity | baseline
  Differences of blood LRRK2 activity measured by the optimized laboratory protocols among LRRK2 G2385R carriers and non-carriers with or without PD
Immune function | baseline
  Immune-related differences between LRRK2 G2385R carriers and non-carriers with or without PD. Immunological measures include (a) distribution of peripheral blood lymphocyte populations: flow cytometry analysis for surface staining of CD19, CD22, CD79A, PAX5 on B cells, and CD11b, CD14, CD16 on monocytes; (b) cytokine profiles in serum: IL-6, IFN-γ, TGF-β, TNF-α; (c) flow cytometry analysis for proteins involved in several LRRK2-related immune signaling pathways: TLR-4, IFN-γ and TGF-β, NF-κB.

SECONDARY OUTCOMES:
Clinical symptoms associated with blood LRRK2 activity | baseline
  Non-motor and motor symptoms are measured using the following methods: Brief Smell Identification Test (B-SIT) , Hamilton Depression Rating Scale (HAM-D) , RBD Questionnaire-Hong Kong (RBDQ-HK), Mini-Mental State Examination (MMSE), Non-Motor Symptoms Scale for Parkinson's Disease (NMSS), MDS-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) and Purdue Pegboard

CONTACTS AND LOCATIONS:
Overall Officials: Piu Chan, MD, PhD, Principal Investigator — Xuanwu Hospital of Capital Medical University
Locations (1):
- Xuanwu Hospital of Capital Medical University, Beijing, China